CLINICAL TRIAL: NCT02529345
Title: CLEAR-ROAD; a Physician-initiated Carotid Trial Investigating the Efficacy of Endovascular Treatment of Carotid Arterial Disease With the Multi-layer RoadSaver Stent
Brief Title: Clear-Road Trial, Investigating the Efficacy of the RoadSaver Stent
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-130919
Record Dates: First submitted 2015-04-27; First posted 2015-08-20 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RoadSaver stent (Experimental): patient treated with the RoadSaver stent of Terumo
  Interventions: Device: RoadSaver stent

INTERVENTIONS:
Device: RoadSaver stent — lesion treated with RoadSaver stent of Terumo

SUMMARY:
The objective of this clinical investigation is to evaluate the clinical outcome (up to 12 months) of treatment by means of stenting with the RoadSaver (Terumo) in subjects at high risk for carotid endarterectomy requiring carotid revascularization due to significant extra-cranial carotid artery stenosis.

DETAILED DESCRIPTION:
It is a Prospective, multi-center, physician-sponsored clinical study.

The objective of this clinical investigation is to evaluate the clinical outcome (up to 12 months) of treatment by means of stenting with the RoadSaver (Terumo) in subjects at high risk for carotid endarterectomy requiring carotid revascularization due to significant extra-cranial carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

High risk for carotid endarterectomy due to anatomical or co-morbid conditions and either:

* has neurological symptoms and ≥ 50% stenosis via angiography, or
* is asymptomatic and has ≥ 80% stenosis via angiography.

  1. Target lesion located in the distal common carotid artery (CCA), internal carotid artery (ICA), or carotid bifurcation.
  2. Arterial segment to be stented has a diameter between 4mm and 9mm
  3. Age ≥ 18 years.
  4. Life expectancy > 12 months from the date of the index procedure.
  5. Provides a signed, IRB (Institutional Review Board) / IEC (Institutional Ethical Committee) approved informed consent form prior to participation.
  6. Willing and able to comply with follow-up requirements.

Exclusion Criteria:

1. Contra-indication to percutaneous transluminal angioplasty (PTA).
2. Sever vascular tortuosity or anatomy that would preclude the safe introduction of a guide catheter, sheath, embolic protection system or stent system.
3. Lesions in the ostium of the common carotid artery.
4. Occlusion of the target vessel.
5. Evidence of intraluminal thrombus.
6. Known sensitivity to nickel-titanium.
7. Known allergy to heparin, aspirin or other anticoagulant/antiplatelet therapies, or is unable or unwilling to tolerate such therapies.
8. Uncorrectable bleeding disorders, or will refuse block transfusion.
9. History of prior life-threatening contrast media reaction.
10. Previous stent placement in the target vessel.
11. Evolving stroke or intracranial haemorrhage.
12. Previous intracranial haemorrhage or brain surgery within the past 12 months.
13. Clinical condition that makes endovascular therapy impossible or hazardous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
30-day rate of Major Adverse events (MAE) | 30 days
  The primary endpoint of this study is the 30-day rate of major adverse events (MAE), defined as the cumulative incidence of any peri-procedural (≤ 30 days post-procedure) death, stroke or myocardial infarction (MI).

SECONDARY OUTCOMES:
Late Ipsilateral stroke | day 31 through 365 days
  number of patients presenting late ipsilateral stroke within day 31 through 365 days
System Technical Success | procedure (day 0)
  Defined as the ability to cross and stent the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex imaging.
device malfunctions | procedure (day 0)
  number of device malfunctions during procedure
Major Adverse Events (MAE's) | at 1,6 and 12 month follow-up
  number of MAE's at the different time frames
serious device-related and procedure-related Adverse Events (SAE's) | at 1, 6 and 12 month follow-up
  number of SAE's at the different time frames
freedom from Target Lesion Revascularization (TLR) | at 1, 6 and 12-month follow-up
  Defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal an distal to the treated lesion edge.
in-stent restenosis (ISR) | at 1, 6 and 12 month follow-up
  patients representing ISR at the different time frames

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — A.Z. Sint-Blasius Hospital
Locations (4):
- Belgium (4):
  - Imelda Hospital, Bonheiden, Antwerp
  - OLV Aalst, Aalst, Oost-Vlaanderen
  - AZ Sint-Blasius, Dendermonde, Oost-Vlaanderen
  - RZ Heilig Hart Hospital, Tienen